CLINICAL TRIAL: NCT07279675
Title: Clinical Predictors of Severity in Pediatric Community-Acquired Pneumonia at Assiut University Children's Hospital
Acronym: CAP-Severity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Sayed Hassan, Resident, Pediatrics, Assiut University
Other Study IDs: AUC-PEDE-CAP-2025
Record Dates: First submitted 2025-11-27; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Community-Acquired Pneumonia; Pediatric Pneumonia; Lower Respiratory Tract Infection
Keywords: Community-acquired pneumonia; Clinical risk factors; Hypoxemia
MeSH Terms: conditions — Community-Acquired Pneumonia; Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children With Community-Acquired Pneumonia: This cohort includes all children aged 1 month to 5 years diagnosed with community-acquired pneumonia (CAP) who present to the pediatric emergency department or are admitted to the pediatric wards of Assiut University Children Hospital during the study period (October 2025 - October 2026).
  All participants will undergo systematic assessment of severity using clinical predictors, laboratory tests, radiological imaging, and the Respiratory Index of Severity in Children (RISC) score.
  Interventions: Other: Assessment of Pneumonia Severity

INTERVENTIONS:
Other: Assessment of Pneumonia Severity — Participants undergo structured evaluation for pneumonia severity, including:
  Clinical predictors (respiratory rate, chest indrawing, hypoxemia, feeding difficulty, mental status, comorbidities) Laboratory markers (complete blood count, RDW, CRP, HCO₃-) Radiological assessment (chest X-ray, CT if indicated) Calculation of RISC score

SUMMARY:
This study aims to identify the clinical factors that predict the severity of community-acquired pneumonia (CAP) in pediatric patients. Children admitted to Assiut University Children's Hospital with a diagnosis of CAP will be evaluated through clinical examination, vital signs, laboratory investigations, and radiological findings. The study focuses on determining which clinical features are associated with more severe disease, higher need for oxygen therapy, intensive care admission, or complications. Understanding these predictors may help clinicians recognize severe cases earlier and improve patient management and outcomes.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is one of the most common causes of morbidity and hospitalization among children worldwide. Early recognition of severe cases is essential for timely intervention. However, clinical predictors of severity in pediatric CAP vary across populations, and there is a need for locally applicable evidence to guide clinical decision-making.

This observational cross-sectional study will enroll pediatric patients presenting with community-acquired pneumonia to Assiut University Children's Hospital. The diagnosis of CAP will be established based on clinical assessment and radiological confirmation. For each patient, demographic data, presenting symptoms, physical examination findings, vital signs, laboratory investigations, and radiological features will be recorded systematically according to the study protocol.

The primary objective of this study is to identify the clinical and laboratory predictors that are significantly associated with severe pneumonia. Severity will be assessed based on predefined criteria, including oxygen requirement, respiratory distress indicators, complications, and need for intensive care admission. Secondary objectives include describing the distribution of severity levels among the enrolled patients and assessing the relationship between individual risk factors and disease outcomes.

The results of this study are expected to provide clinically relevant predictors that can support early identification of severe CAP in children, improve triage decisions, and optimize treatment strategies within similar healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 5 years.
* Children of both sexes
* Onset of illness in the community, not more than 48 hours after hospital admission.

Exclusion Criteria:

* Children below 1 month, as neonatal pneumonia differs in pathology and management from CAP.
* Children with hospital-acquired pneumonia
* Known primary or secondary immunodeficiency
* Children with chronic respiratory diseases (as cystic fibrosis, bronchiectasis) or congenital lung malformations.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 month to 5 years of both sexes diagnosed with community-acquired pneumonia (CAP) presenting to the pediatric emergency department or admitted to pediatric wards at Assiut University Children's Hospital during the study period (October 2025 - October 2026). Children with hospital-acquired pneumonia, known immunodeficiency, chronic respiratory diseases, or congenital lung malformations are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Association of Severity Scores with Clinical Outcomes | 14 days from enrollment (typical hospital stay and outpatient follow-up)
  The primary outcome will be the correlation coefficient (r value) between the Community-Acquired Pneumonia (CAP) severity score and each clinical outcome.
  The clinical outcomes will include:
  Length of hospital stay (days) Oxygen requirement (L/min) ICU admission (yes/no) Occurrence of complications (yes/no) Mortality (yes/no)
Severity of Community-Acquired Pneumonia Assessed by the Respiratory Index of Severity in Children (RISC) | 4 days from enrollment (typical hospital stay and outpatient follow-up)
  CAP severity will be assessed using the Respiratory Index of Severity in Children (RISC) score.
  The RISC score ranges from 0 to 6, with higher scores indicating more severe disease.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serin O, Akbasli IT, Cetin SB, Koseoglu B, Deveci AF, Ugur MZ, Ozsurekci Y. Predicting Escalation of Care for Childhood Pneumonia Using Machine Learning: Retrospective Analysis and Model Development. JMIRx Med. 2025 Mar 4;6:e57719. doi: 10.2196/57719. PMID 40036666
- [Background] Kapoor A, Awasthi S, Kumar Yadav K. Predicting Mortality and Use of RISC Scoring System in Hospitalized Under-Five Children Due to WHO Defined Severe Community Acquired Pneumonia. J Trop Pediatr. 2022 Jun 6;68(4):fmac050. doi: 10.1093/tropej/fmac050. PMID 35727140
- [Background] Anteneh ZA, Arega HE, Mihretie KM. Validation of risk prediction for outcomes of severe community-acquired pneumonia among under-five children in Amhara region, Northwest Ethiopia. PLoS One. 2023 Feb 15;18(2):e0281209. doi: 10.1371/journal.pone.0281209. eCollection 2023. PMID 36791115
- [Background] O. Shukla, N. Rathwa, and L. Mude, "Assessment of severity of community acquired pneumonia by paediatric infectious diseases society and clinical and radiological profile in 0-5 year age group," 2024, Accessed: Sep. 17, 2025.